CLINICAL TRIAL: NCT00402402
Title: Comparison of Quantiferon-TB Gold Assay With Tuberculin Skin Testing for Detecting Latent Mycobacterium Tuberculosis Infection in Patients With Chronic Liver Disease Awaiting Liver Transplantation
Brief Title: Comparison of Quantiferon-TB Gold Assay With Tuberculin Skin Testing in Patients With Chronic Liver Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 06-0648-AE
Record Dates: First submitted 2006-11-21; First posted 2006-11-22 (Estimated); Last update posted 2008-04-16 (Estimated); Status verified 2006-11

CONDITIONS: Chronic Liver Disease; Liver Transplantation; Tuberculosis
Keywords: Tuberculin skin test; Quantiferon-TB Gold assay; Chronic liver disease; Liver transplantation; Latent tuberculosis infection
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis | interventions — Tuberculin

INTERVENTIONS:
Procedure: Tuberculin skin test
Procedure: Quantiferon-TB Gold assay

SUMMARY:
The purpose of the study is to estimate the usefulness of the QuantiFERON®-TB Gold test for the diagnosis of latent tuberculosis infection in liver transplant candidates by correlating the test results with risk factors for LTBI

DETAILED DESCRIPTION:
Tuberculosis (TB) is an important cause of morbidity and mortality in organ transplant recipients. Although the tuberculin skin test (TST) is recommended for screening of latent tuberculosis infection (LTBI) in all candidates for liver transplantation, the performance of the TST in this setting is less than optimal, due to a lack of specificity and a lack of sensitivity in a population that is relatively immunocompromised. Recently, a new test named QuantiFERON-TB Gold (QFT-G) has been approved for the diagnosis of LTBI. QFT-G is expected to be more specific than TST. However, there are no studies defining the performance of QFT-G in a population of patients on a waiting list for liver transplantation. We plan to estimate the usefulness of the QFT-G test for the diagnosis of LTBI in a cohort of patients with end-stage liver disease. We hypothesize that the QFT-G test will correlate better with the risk of LTBI.

ELIGIBILITY:
Inclusion Criteria:

* Chronic liver disease on the waiting list or being wait listed for liver transplantation

Exclusion Criteria:

* Unable to provide informed consent

  * Previous history of immediate hypersensitivity to TST
  * Previous severe local ulceration with TST
  * Suspected active TB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-10; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Concordance between the Quantiferon-TB Gold assay and the tuberculin skin test
Correlation of the test results to the patient's risk of latent TB infection

SECONDARY OUTCOMES:
Factors associated with discordance between the TST and the QFT-G test
Frequency of anergy in this patient population

CONTACTS AND LOCATIONS:
Overall Officials: Deepali Kumar, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Univcersity Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Background] Benito N, Sued O, Moreno A, Horcajada JP, Gonzalez J, Navasa M, Rimola A. Diagnosis and treatment of latent tuberculosis infection in liver transplant recipients in an endemic area. Transplantation. 2002 Nov 27;74(10):1381-6. doi: 10.1097/00007890-200211270-00006. PMID 12451235
- [Background] Ferrara G, Losi M, Meacci M, Meccugni B, Piro R, Roversi P, Bergamini BM, D'Amico R, Marchegiano P, Rumpianesi F, Fabbri LM, Richeldi L. Routine hospital use of a new commercial whole blood interferon-gamma assay for the diagnosis of tuberculosis infection. Am J Respir Crit Care Med. 2005 Sep 1;172(5):631-5. doi: 10.1164/rccm.200502-196OC. Epub 2005 Jun 16. PMID 15961696
- [Background] Pai M, Gokhale K, Joshi R, Dogra S, Kalantri S, Mendiratta DK, Narang P, Daley CL, Granich RM, Mazurek GH, Reingold AL, Riley LW, Colford JM Jr. Mycobacterium tuberculosis infection in health care workers in rural India: comparison of a whole-blood interferon gamma assay with tuberculin skin testing. JAMA. 2005 Jun 8;293(22):2746-55. doi: 10.1001/jama.293.22.2746. PMID 15941804